CLINICAL TRIAL: NCT05018845
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Chronic Kidney Disease.
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for CKD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-20-ATG-22
Record Dates: First submitted 2021-08-20; First posted 2021-08-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Renal Failure; stem cell treatment; Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Chronic Kidney Disease.

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Chronic Kidney Disease (CKD). This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of CKD. Patients with CKD will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous Effector cells (activated lymphocytes) treatment will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Kidney Disease
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: creatinine levels | Four year follow-up
  It will be completed for each follow up point.
Efficacy: changes in eGFR | Four year follow-up
  It will be completed for each follow up point.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belingheri M, Lazzari L, Parazzi V, Groppali E, Biagi E, Gaipa G, Giordano R, Rastaldi MP, Croci D, Biondi A, Rebulla P, Edefonti A, Ghio L. Allogeneic mesenchymal stem cell infusion for the stabilization of focal segmental glomerulosclerosis. Biologicals. 2013 Nov;41(6):439-45. doi: 10.1016/j.biologicals.2013.09.004. Epub 2013 Oct 14. PMID 24135082
- [Background] Rahyussalim AJ, Saleh I, Kurniawati T, Lutfi APWY. Improvement of renal function after human umbilical cord mesenchymal stem cell treatment on chronic renal failure and thoracic spinal cord entrapment: a case report. J Med Case Rep. 2017 Nov 30;11(1):334. doi: 10.1186/s13256-017-1489-7. PMID 29187247